CLINICAL TRIAL: NCT04391608
Title: Randomized Trial of Tenofovir Disoproxil Fumerate Dose Adjustment VS. Switching to Tenofovir Alafenamide in Tenofovir Disoproxil Fumarate-experienced Chronic Hepatitis B Patients With Renal Impairment
Brief Title: TDF Dose Adjustment VS. Switching to TAF in TDF-experienced CHB Patients With Renal Impairment
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Watcharasak Chotiyaputta, Associate professor, Faculty of Medicine, Siriraj Hospital, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Si 798/2019
Record Dates: First submitted 2020-05-06; First posted 2020-05-18 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-03

CONDITIONS: Renal Insufficiency; Tenofovir
Keywords: Tenofovir; Tenofovir disoproxil fumarate; Tenofovir alafenamide; TDF; TAF; Renal; Impairment; Insufficiency
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tenofovir Alafenamide (Active Comparator): Tenofovir Alafenamide 25 mg/day
  Interventions: Drug: Switching to Tenofovir Alafenamide
- TDF dose reduction (No Intervention): TDF dose reduction

INTERVENTIONS:
Drug: Switching to Tenofovir Alafenamide — Switching from Tenofovir Disoproxil Fumarate to Tenofovir Alafenamide
  Other Names: Switching from Tenofovir Disoproxil Fumarate to Tenofovir Alafenamide
  Arms: Tenofovir Alafenamide

SUMMARY:
Tenofovir is a nucleotide analog drug that works against both Human immunodeficiency virus (HIV) and HBV. TDF and TAF are prodrug of Tenofovir. TAF has a higher plasma stability than TDF, which makes TDF require a higher dose to get the concentration of drugs in the liver equal to the amount of TAF.

Previous studies have shown the effects of TAF once daily and TDF once daily on kidney function and bone mass. The efficacy of TAF in virus suppression is comparable to TDF, but the effect on the kidneys and bone mass from TAF has less side effects than TDF. In addition, changing the medication from TDF to TAF shows that kidney function tends to improve.

Hepatitis B patients taking TDF have adjusted their dosage due to impair renal function, for example, from 1 time per day to every 48 hours or every 72 hours. This group of patients does not have a clear evidence-based recommendation for choosing a reduced dose of TDF or change to TAF. Therefore, the main objective of this study is to study patients with hepatitis B who have taken TDF and have renal function impairment that have been adjusted. Taking the same medicine with dose adjustment or changing the drug to TAF which treatment will more improve the kidney function.

DETAILED DESCRIPTION:
Hepatitis B virus is a global public health problem. More than 250 million people are infected worldwide. These infections lead to chronic hepatitis, cirrhosis and liver cancer. According to past statistics, infection with hepatitis B virus is an important factor of death in 880,000 patients per year.

Patients who receiving natural immunity or receiving antiretroviral therapy that loss of hepatitis B surface antigen (HBsAg loss) reduce the risk of cirrhosis and hepatocellular carcinoma (HCC). HBsAg loss is now considered the target of treatment.

Nucleot(s)ide is an antiviral drug that can reduce the number of viruses, reduce the risk of HCC and death from Hepatitis B viral infection. The most widely used drugs are Lamivudine (LMV), Entecavir (ETV), Tenofovir disoproxil fumerate (TDF) and Tenofovir alafenamide (TAF). However, Nucleotide is unable to eliminate the Hepatitis B virus from the liver cells of the infected person due to covalently closed. circular DNA (cccDNA), which is a template for viral replication. Therefore, long-term Nucleotide therapy is necessary. As a result, patients may have side effects from the treatment when taking medication for a long time, such as viral resistance in Lamivudine, deterioration of kidney function and osteoporosis in Tenofovir.

Tenofovir is a nucleotide analog drug that works against both Human immunodeficiency virus (HIV) and HBV. TDF and TAF are prodrug of Tenofovir. TAF has a higher plasma stability than TDF, which makes TDF require a higher dose to get the concentration of drugs in the liver equal to the amount of TAF.

The side effects of Tenofovir treatment found on the kidneys and bones which are problems for long-term treatment. It is recommended to reduce the dose of TDF in patients with renal function reduced to less than 50 ml / min as shown in Table but do not have to adjust the dose of TAF except when the GFR value is less than 15 ml / min. it is recommended to stop taking TAF if severe renal impairment.

Previous studies have shown the effects of TAF once daily and TDF once daily on kidney function and bone mass. The efficacy of TAF in virus suppression is comparable to TDF, but the effect on the kidneys and bone mass from TAF has less side effects than TDF. In addition, changing the medication from TDF to TAF shows that kidney function tends to improve. Therefore, there is a recommendation in the practice guideline to change from TDF to TAF or ETV in patients who use TDF and there is a risk of kidney problems or thin bone mass based on history for LMV resistance (if LMV resistance, ETV should not be used because HBV is more resistant to ETV).

Hepatitis B patients taking TDF have adjusted their dosage due to impair renal function, for example, from 1 time per day to every 48 hours or every 72 hours. This group of patients does not have a clear evidence-based recommendation for choosing a reduced dose of TDF or change to TAF. Therefore, the main objective of this study is to study patients with hepatitis B who have taken TDF and have renal function impairment that have been adjusted. Taking the same medicine with dose adjustment or changing the drug to TAF which treatment will more improve the kidney function.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 - 75 years old
2. Chronic hepatitis B virus infection
3. Reduced renal function and need to adjust the dose of TDF
4. Have an eGFR of > 15 ml / min.
5. HBV DNA viral load levels < 10 U/mL in the last 3 months before participating in the project
6. No HCC by Ultrasonography of the upper abdomen or CT 3-phase of liver or MRI liver in the 3 months before participating in the project.

Exclusion Criteria:

1. HIV infection or hepatitis C or hepatitis D co-infection
2. Decompensated cirrhosis, including variceal bleeding, ascites, hepatic encephalopathy
3. Active hepatocellular carcinoma or during the 3 years after treatment
4. Solid organ transplantation or Bone marrow transplantation
5. Chronic kidney disease caused by glomerulonephritis, tubulo-interstitial nephritis), Obstructive uropathy or autosomal dominant polycystic kidney, and Kidney disease from other causes
6. Diabetes with HbA1c> 8 or uncontrollable hypertension
7. Active malignancy of cancer in other organs in the last 3 years
8. History of receiving non-steroidal anti-inflammatory drugs (NSAIDs) or other nephrotoxic drugs within the past 1 month (except tenofovir) (For patients receiving NSAIDS after participating in this study, patients were advised to stop taking NSAIDs but not exclude from the study)
9. Receive immunosuppressive drug
10. Pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-11-09 (Actual); Primary Completion 2022-07-31 (Estimated); Study Completion 2022-07-31 (Estimated)

PRIMARY OUTCOMES:
Renal safety assessed by changes in eGFR | 48 weeks
  To study renal function changes by measuring eGFR during Tenofovir disoproxil fumarate (TDF) dose reduction versus switching to Tenofovir alafenamide (TAF) after 48 weeks of treatment in chronic hepatitis B with impaired kidney function

SECONDARY OUTCOMES:
Renal safety assessed by changes in urine sugar (0 to 4+) | 48 weeks
  To study kidney function changes by measuring urine sugar (0 to 4+) during TDF dose reduction compared to switching to TAF after 48 weeks of treatment
Renal safety assessed by changes in urine protein creatinine ratio | 48 weeks
  To study kidney function changes by measuring urine protein creatinine ratio during TDF dose reduction compared to switching to TAF after 48 weeks of treatment
Renal safety assessed by changes in urine ß2-microglobulin (µg/mL) | 48 weeks
  To study kidney function changes by measuring urine ß2-microglobulin (µg/mL) during TDF dose reduction compared to switching to TAF after 48 weeks of treatment
Renal safety assessed by changes in urine phosphate (mg/dL) | 48 weeks
  To study kidney function changes by measuring urine phosphate(mg/dL) during TDF dose reduction compared to switching to TAF after 48 weeks of treatment
Renal safety assessed by changes in urine neutrophil gelatinase-associated lipocalin (NGAL) (ng/mL) | 48 weeks
  To study kidney function changes by measuring urine neutrophil gelatinase-associated lipocalin (NGAL) (ng/mL) during TDF dose reduction compared to switching to TAF after 48 weeks of treatment
Efficacy of viral suppression assessed by amount of hepatitis B (HBV DNA) (IU/mL) | 48 weeks
  To study the efficacy of treatment by measuring amount of hepatitis B (HBV DNA) (IU/mL) during the dose reduction of TDF compared to switching to TAF after 48 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Watcharasak Chotiyaputta, Asso Prof, Principal Investigator — Mahidol University
Locations (1):
- Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkok Noi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-25): https://cdn.clinicaltrials.gov/large-docs/08/NCT04391608/Prot_SAP_002.pdf